CLINICAL TRIAL: NCT04923633
Title: The Reproducibility and Consistency of Instrument-assisted Soft Tissue Manipulation
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary T. Loghmani, Associate Professor, Indiana University
Other Study IDs: 10329; R41AT011494 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-06-11 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Massage
Keywords: Soft tissue manipulation, massage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Phase I Instrument-Assisted Soft Tissue Manipulation (IASTM) Stroke Pattern Analysis: Fifteen (n=15) experienced clinicians, each with 8 or more years experiences in instrument-assisted soft tissue manipulation (IASTM), will participate in an observational studying analyzing their application of basic stroke patterns (linear, curved) to a consistent research assistant/model. IASTM is a type of massage that uses rigid devices. A Quantifiable Soft Tissue Manipulation (QSTM) device system will be used for determining objective metrics of stroke parameters (e.g. stroke force, rate, angle) and results will be compared between participants to determine characteristic stroke profile patterns for use in training and research.
- Phase II Consistency of IASTM Force Application: The reproducibility of applying a targeted STM stroke force will be determined within and between therapists, both with and without visual monitoring of the QSTM metrics and graphic display. Two novice and two experienced therapists will be trained using QSTM. A novice is defined as a clinician with <1 year and an experienced with >8 years of practice. Fifty (n=50) healthy, non-obese subjects will be enrolled that meet the inclusion/exclusion criteria. First, the clinicians will apply a self-perceived "moderate" force for 15sec (non-therapeutic dose), within subject tolerance, without using QSTM feedback. Then, the clinician will apply a targeted force of 10N with visual monitoring of QSTM feedback. This process will be repeated 5-7 days later to determine repeatability. After testing, subjects will participate in simple back and/or leg stretches and an ice pack applied.
- Phase III Reliability of Dynamic Pressure Pain Threshold Assessment: The reliability of dynamic pressure pain threshold (DPPT) assessment over a specified area will be determined. Two novice and two experienced clinicians will be trained using QSTM. Subjects (n=50) will be recruited that meet the inclusion/exclusion criteria of healthy, non-obese, younger (≥18 but ≤30yo) and older individuals (≥50 but ≤75yo) (males and females). The clinicians will apply force to standardized areas of the back and thigh regions for 1 min, using the Quantifiable Soft Tissue Manipulation (QSTM) device system. The force applied will be applied up to but below the threshold of when a subject says to "stop" when they feel the "pressure" change into any sort of "irritating discomfort/pain." Secondary clinical outcomes will be assessed before and after testing since testing could have effects on the soft tissue, pain, and physical performance measures. After testing, the subject will be instructed in simple back and/or leg stretches and an ice pack applied.
  Interventions: Device: Quantifiable Soft Tissue Manipulation (QSTM)

INTERVENTIONS:
Device: Quantifiable Soft Tissue Manipulation (QSTM) — Quantifiable soft tissue manipulation (QSTM) is a force sensing device system that can be used by a clinician to apply a massaging force while the system monitors objective metrics, i.e., the amount, rate, and angle of force applied.
  Groups: Phase III Reliability of Dynamic Pressure Pain Threshold Assessment

SUMMARY:
The overall purpose of this study is to objectively describe and test the consistency and reproducibility of instrument-assisted soft tissue manipulation (IASTM).The specific aims of this current study are to:

1. Analyze IASTM stroke patterns using objective metrics;
2. Test the consistency of force application, with and without visual monitoring of objective metrics, and;
3. Determine the reliability of dynamic pressure pain threshold assessment. The ultimate goal of this continuing line of research is to improve soft tissue manual therapy practice in research, education, and clinic for use as a non-invasive modality in soft tissue assessment and treatment. Results from this protocol will inform future clinical trials, including studies exploring the effects of different IASTM dose-loads in various musculoskeletal pain conditions.

DETAILED DESCRIPTION:
This is a single-site study consisting of three study phases. Phase I will observe and analyze clinician's application of instrument-assisted soft tissue manipulation (IASTM) as a means to identify signature profiles for the stroke rate, angle, and direction that are characteristic of basic (e.g., linear, curved) stroke patterns. Phase II will assess the consistency of IASTM force application. Phase III will assess the reliability of dynamic pressure pain threshold assessment. Clinician participants (Phase I) will attend one study visit consisting of basic linear and curved IASTM stroke pattern applications and complete a questionnaire. Total study duration for clinician participants will be 90 minutes. Non-clinician subjects will attend two study visits (Phase II) or one study visit (Phase III). Visits will consist of completion of questionnaires, application of IASTM strokes by a clinician using the QSTM device, and stretching.

ELIGIBILITY:
Inclusion Criteria:

Phase I

1. Male or female between the ages of 18-75 years old.
2. Be a licensed, practicing healthcare clinician (e.g. physical therapist, massage therapist, osteopathic physician, athletic trainer, chiropractor)
3. Have at least 8 years of clinical experience in instrument-assisted soft tissue manual therapy

Phase II

1. Male and female subjects between 18-75 years old
2. Body Mass Index (BMI) ≥ 18.5 kg/m2 but <30 kg/m2

Phase III

1. Male and female subjects, ages younger (≥18 but ≤30yo) and older (≥50 but ≤75yo)
2. Body Mass Index (BMI) ≥ 18.5 kg/m2 but <30 kg/m2

Exclusion Criteria:

Phase I

1. <8 years of clinical experience in instrument-assisted soft tissue manual therapy practice
2. Any known pain conditions, such as nerve impingement (radiculopathies), rheumatoid arthritis, osteoarthritis, or any other inflammatory conditions that could interfere with the participant's ability to perform basic IASTM stroke patterns.
3. Any known cardiovascular, pulmonary, or metabolic disease that could interfere with the clinician's ability to perform basic IASTM stroke patterns.

Phase II

1. Known cardiovascular, pulmonary, or metabolic disease;
2. Current smoking or those who quit smoking within the previous 6 months;
3. Current use of anti-inflammatory or analgesics;
4. Any history of back, neck, lower extremity, or abdominal surgery or injury; or back, neck, or leg pain within the previous 6 months that impaired function;
5. Any co-morbidities that could contribute to back, neck, or leg pain (e.g., radiculopathies, rheumatoid arthritis, osteoarthritis, inflammatory conditions).

Phase III 1. The same exclusion criteria as for Phase II.

-

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy, males and females, ages 18-75.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Phase I Stroke Pattern Characteristic Descriptions | Analysis results within 6 months.
  The objectives metrics from quantifiable soft tissue manipulation device system will be analyzed for common or characteristic applications between clinicians.
Phase II Reliability of IASTM Force Application | Measured within 2 hours for same day reliability and at 7 days for between day reliability. Results reported by end of study at one year
  The agreement in soft tissue manipulation force application, between and within clinicians, will be determined within a single session and between session (within 7 days apart).
Phase III Reliability of Dynamic Pressure Pain Threshold Assessment | Measured within 2 hours on same day of testing. Results reported by end of study at one year.
  The agreement between and within clinicians in pressure pain threshold assessment over a body area will be determined within a single session.

SECONDARY OUTCOMES:
(Phase III Only) Heart Rate | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Radial pulse will be palpated to determine heart rate (in beats per minute, BPM).
(Phase III Only) Blood Pressure | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Will determine systolic and diastolic blood pressure (in mmHg) using a stethoscope and sphygmomanometer.
(Phase III Only) Range of Motion | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Will measure the amount (range) of trunk movement (in degrees) using a modified protractor.
(Phase III Only) Hamstring Length Flexibility Test. | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Will measure the amount (range) of passive knee extension movement available (in degrees) with the hip stabilized at 90 degrees using a modified protractor.
(Phase III Only) Trunk Forward Bend Flexibility Test. | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  A tape measurer/ruler will be used to determine the extensibility (e.g. limberness) of the posterior (back) trunk soft tissues during seated trunk forward bend (reaching) muscle length test (change from start to end of test measured in centimeters).
(Phase III Only) Strength | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  A handheld dynamometer will be used to test the strength (Newtons of force) of the subject's back and thigh.
(Phase III Only) Static Pressure Pain Threshold | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  This test will determine a subject's pressure pain sensitivity in a single spot using a non-invasive device, i.e. static algometer.
(Phase III Only) Skin Surface Temperature | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Changes in skin surface temperature will be determined using an infrared thermometer of the skin are where IASTM is applied on the back and thigh.
(Phase III Only) 10-Meter Walk Test (10-MWT) | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  Maximal walking speed (MWS) (in meters/sec) will be determined using the 10-meter walk test as a functional performance measure.
(Phase III Only) Vertical Jump Test | Measured before and within 2 hours after IASTM force application. Results reported by end of study at one year.
  The vertical jumping height (in centimeters) (only in subjects 18-30 y.o.) will be determined as a functional performance measure

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Loghmani, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After July 31, 2022 for one year
Access Criteria: Other research institution PI or as requested upon review.